CLINICAL TRIAL: NCT05223816
Title: An Open-Label, Multiple-Center, Phase IIa/IIb Clinical Trial to Evaluate the Efficacy, Safety and Tolerability of VG161 as Monotherapy and in Combination With Nivolumab for Treatment of Patients With Hepatocellular Carcinoma or Intrahepatic Cholangiocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Virogin Biotech Canada Ltd (Industry)
Responsible Party: Sponsor
Organization: Virogin Biotech Ltd. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VG161-A201
Record Dates: First submitted 2021-12-20; First posted 2022-02-04 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Hepatocellular Carcinoma; Intrahepatic Cholangiocarcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular; Cholangiocarcinoma | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Safety Run-in Cohort (Experimental): 10 patients will be treated with IT injection of VG161 in the cohort 1 at dose level of 1.0x10E8 PFU x 3 days.
  Interventions: Drug: VG161
- Cohort 2 (HCC) (Experimental): 21 patients will be treated with IT injection of VG161 in the cohort 1 at dose level of 1.0x10E8 PFU x 3 days.
  Interventions: Drug: VG161
- Cohort 3 (ICC) (Experimental): 20 patients will be treated with IT injection of VG161 in the cohort 1 at dose level of 1.0x10E8 PFU x 3 days.
  Interventions: Drug: VG161
- Cohort 4 (HCC and ICC) (Experimental): Up to 12 patients will be treated with IT injection of VG161 ar dose level of 1.0x10E8 PFU x 3 days. and Nivolumab per approved label.
  Interventions: Drug: VG161; Drug: Nivolumab Injection [Opdivo]

INTERVENTIONS:
Drug: VG161 — Name: VG161 (Recombinant Human IL12/15-PDL1B Oncolytic HSV-1 Injection (Vero Cell)) Concentration/Content: ≥1×107 PFU/mL; 1.0 mL/vial. Actual titer will be recorded on Certificate of Analysis.
  Composition: VG161,50 mM Tris-HCl, 150mM NaCl, <5% glycerol Route of Administration: Intratumoral injection or image guided intratumoral injections.
Drug: Nivolumab Injection [Opdivo] — immunotherapy treatment
  Arms: Cohort 4 (HCC and ICC)

SUMMARY:
Safety Run-in Cohort (cohort 1):

10 patients will be treated with IT injection of VG161 in the cohort 1 at dose level of 1.0x10E8 PFU x 3 days.

Monotherapy Cohorts (Cohort 2 and 3) Cohort 2 (HCC) This part is a single-agent, single one-dose level and single-arm design. Approximately 39 subjects will be enrolled in the study to receive VG161. In the first stage, 21 subjects will be enrolled. If there is only 1 or fewer subjects has been observed with objective response and no more than 12 (<13) subjects have PFS longer than 3 months, the trial will be stopped. Otherwise, this study will continue to enter the second stage, and 18 additional subjects will be added, and the total number of trial subjects will reach 39.

Cohort 3 (ICC) This part is a single-agent, single one-dose level and single-arm design. The trial will be carried out in two periods. In the first period, a total of 20 subjects will be enrolled. If there is only 1 or fewer response case in the 20 subjects, the trial will be stopped to investigate the efficacy of the IP, otherwise, subjects will continue to enter the second period, and 13 additional subjects will be added, and the total number of trial cases will reach 33.

Cohort 4 (ICC and HCC) Combination with Nivolumab Combination cohort and subjects will receive VG161 at the same schedule as the monotherapy cohorts and 240 mg of intravenous Nivolumab on days 8 and 15 of each treatment cycle. The Nivolumab dose can be changed to 480 mg every 4 weeks after cycle one based on investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent.
2. Males or females aged 18 years and older.
3. Performance status: Eastern Cooperative Oncology Group (ECOG) 0 or 1.
4. For subject in Cohort 2: cytologically confirmed advanced/metastatic or surgically unresectable HCC, with documented disease progression after at least two lines of FDA approved systemic therapy, including immunotherapy or anti-angiogenesis therapy as the first line treatment and at least one regimen of the following agents as the second line: anti-angiogenesis agents, tyrosine kinase inhibitors or immunotherapy.
5. For subject in Cohort 3: Histologically or cytologically confirmed advanced/metastatic or surgically unresectable ICC, with documented disease progression after chemotherapy as the first line systemic therapy. For patients with known IDH1 mutation, they must receive the appropriate targeted therapy with a IDH1 inhibitor and for patients with MSI-H tumors, they must receive immunotherapy with PD-1 inhibitors.
6. For subjects in Cohort 1 and Cohort 4: should fulfill either inclusion criteria 4) or 5).
7. Liver function: Child-Pugh A-B for cohort 1 and 2.
8. At least one measurable lesion per RECIST 1.1
9. At least 1 injectable lesion; ≥15 mm in longest diameter and deemed injectable as per Investigator's discretion. Subjects with deep or visceral lesions (such as hepatic or intraperitoneal lymph nodes) that can be safely injected under guided imaging can be considered for intratumoral injection of VG161..

Exclusion Criteria:

1. Participation in any trial of any other investigational agent within the last 4 weeks prior to dosing. Wash out periods to be reviewed on a case by case basis with Medical Monitor, as required.
2. Tumors to be injected lying in mucosal regions or close to an airway, major blood vessel or spinal cord that, in the opinion of the Investigators, could cause occlusion or compression in the case of tumor swelling or erosion into a major vessel in the case of necrosis.
3. Subjects with any primary Central Nervous System (CNS) malignancy including glioma and current, active, progressing CNS malignancy, including carcinomatosis meningitis are excluded. Subjects with treated brain metastases are eligible if there is no evidence of progression for at least 4 weeks after CNS-directed treatment, as ascertained by clinical examination and brain imaging (magnetic resonance imaging [MRI] or computed tomography [CT] scan) during the screening period and off steroids (for at least 2 weeks prior to first dose of IP).
4. Major surgery within 14 days prior to dosing.
5. Intercurrent serious infections within 28 days prior to Screening or treated systematically with antibiotics within 14 days prior to signing ICF.
6. Life-threatening illness unrelated to cancer.
7. Active Herpes infection.
8. Treatment with antiviral agents within 14 days prior to dosing.
9. Uncontrolled congestive heart failure.
10. Known to test positive for human immunodeficiency virus (HIV) or syphilis.
11. Active infection including hepatitis B (HBV) or hepatitis C (HCV) that currently under anti-virus treatment which can affect study drug treatment as per investigator's decision.
12. Use of ganciclovir or acyclovir within 14 days prior to dosing.
13. Subjects with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days prior to dosing. Inhaled or topical steroids, and adrenal replacement steroid doses ≤10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
14. Subjects who have been on systemic anticoagulants within 14 days prior to dosing and/or with International Normalized Ratio (INR) > 1.5 x the upper limit of the reference range are excluded from this study.
15. Subjects with prior radiation therapy to the tumor lesion to be injected are excluded from the study, unless there is evidence of tumor progression in the most recent imaging, following completion of radiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety in Cohort1 | 12 months
  Occurrence and severity of AEs, SAEs (according to NCI CTCAE version 5.0) in Safety Run-in Cohort (cohort 1)
ORR | 12 months
  Objective response rate in HCC Cohort (Cohort 2) and ICC Cohort (Cohort 3)
PFS | 3 months
  Progression-free survival in HCC Cohort (Cohort 2)

SECONDARY OUTCOMES:
Blood concentration of VG161 | 12 months
  Quantity of Blood concentration of VG161 in cohort 1
PD-L1 blocking peptide and IL12, IL-15 concentrations | 12 months
  Quantity of PD-L1 blocking peptide and IL12, IL-15 concentrations in cohort 1
serum antibodies in cohort 1 | 12 months
  Quantity of serum antibodies in cohort 1
Viral shedding | 12 months
  VG161 DNA tested in cohort 1
Immunogenicity endpoints | 12 months
  serum antibodies (ADA and Nab) at different time points in cohort 1
ORR in cohort 1 | 12 months
  objective response rate in Cohort1
PFS | 12 months
  Progression-free survival in all cohorts
OS | 12 months
  Overall survival rate in all cohorts
DOR | 12 months
  Duration of response in all cohorts
Safety in Cohort2 and Cohort3 | 12 months
  Occurrence and severity of AEs, SAEs (according to NCI CTCAE version 5.0) in cohort 2 and cohort 3
peripheral blood lymphocyte subsets | 12 months
  Quantity of peripheral blood lymphocyte subsets (CD3+, CD4+, CD8+, CD4+/CD8+ ratio, CD19+, CD16+CD56+ (NK) cells) in cohort 2 and cohort 3
plasma cytokines | 12 months
  Quantity of plasma cytokines (IL-15, IL-6, TNF-a, IFN-γ) in cohort 2 and cohort 3
immune-related indicators | 12 months
  Quantity of immune-related indicators (PD-L1, PD-1, CD69, CD8+Ki67high) in cohort 2 and cohort 3
anti-HSV-1 antibody | 12 months
  Quantity of anti-HSV-1 antibody in cohort 2 and cohort 3

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Mayo Clinic, Phoenix, Arizona
  - Mayo Clinic Florida, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- See also: Virogin Biotech Website — https://virogin.com/